CLINICAL TRIAL: NCT00645177
Title: A Phase 2 Randomized, Placebo-Controlled, Double-Blind Study of ABT-869 in Combination With Paclitaxel Versus Paclitaxel Alone as First-line Treatment in Subjects With Locally Recurrent or Metastatic Breast Cancer
Brief Title: Phase 2 Study of ABT-869 in Combination With Paclitaxel Versus Paclitaxel Alone to Treat Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M10-265; 2007-005905-23 (EudraCT Number)
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — linifanib; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Active Comparator): In study, this arm is a randomized (blinded) to ABT-869 arm plus paclitaxel.
  Note: Prior to randomization, approximately 6-12 subjects will be enrolled in open-label lead-in to assess the tolerability of the combination. The initial open-label, lead-in cohort of six subjects will be monitored for 2 cycles (8 weeks) to assess the PK interactions and the safety of the combination of 0.20 mg/kg QD ABT-869 and paclitaxel (90 mg/m2). Enrollment into the randomized portion will begin after a cohort has completed two cycles (8 weeks) of therapy and no toxicities prohibit the cohort from continuing on to Cycle 3.
  Alternative doses may be explored based on the tolerability of the combination
  Interventions: Drug: ABT-869; Drug: paclitaxel
- B (Placebo Comparator): In study, this arm is a randomized (blinded) to placebo for ABT-869 plus paclitaxel arm.
  Note: Prior to randomization, approximately 6-12 subjects will be enrolled in open-label lead-in to assess the tolerability of the combination. The initial open-label, lead-in cohort of six subjects will be monitored for 2 cycles (8 weeks) to assess the PK interactions and the safety of the combination of 0.20 mg/kg QD ABT-869 and paclitaxel (90 mg/m2). Enrollment into the randomized portion will begin after a cohort has completed two cycles (8 weeks) of therapy and no toxicities prohibit the cohort from continuing on to Cycle 3.
  Alternative doses may be explored based on the tolerability of the combination
  Interventions: Drug: paclitaxel; Drug: Placebo for ABT-869

INTERVENTIONS:
Drug: ABT-869 — 0.20 mg/kg (or dose from Lead-in) QD, tablets taken orally days 1-28 of every 28-day cycle
  Arms: A
Drug: paclitaxel — 90 mg/m2 IV infusion over 1 hour, weekly every 3 out of 4 weeks
Drug: Placebo for ABT-869 — 0.20 mg/kg (or dose from Lead-in) QD, tablets taken orally days 1-28 of every 28-day cycle
  Arms: B

SUMMARY:
The purpose of this study is to determine the effect of ABT-869 plus paclitaxel compared to paclitaxel alone on disease progression in metastatic breast cancer.

DETAILED DESCRIPTION:
Only the open-label lead-in portion of the study was enrolled (n=10). The randomized portion was not initiated. N = approximately 102 (90 randomized in a 1:1 ratio in Phase 2, approximately 6-12 enrolled in open-label lead-in to assess the tolerability of the combination) Phase 2, randomized, placebo-controlled, double-blind, multi-center study of the efficacy and tolerability of the ABT-869 + paclitaxel versus placebo for ABT-869 + paclitaxel in subjects with documented metastatic breast cancer in the first line metastatic therapy setting. An initial open-label, lead-in cohort of six subjects will be monitored for 2 cycles (8 weeks) to assess the PK interactions and the safety of the combination of 0.20 mg/kg QD ABT-869 and paclitaxel (90 mg/m2). Enrollment into the randomized portion will begin after a cohort has completed two cycles (8 weeks) of therapy and no toxicities prohibit the cohort from continuing on to Cycle 3. Alternative doses may be explored based on the tolerability of the combination.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be female and > 18 years of age.
* Subject must be diagnosed with adenocarcinoma of the breast.
* Subject must have metastatic disease or locally recurrent disease that is not amenable to surgical resection with curative intent.
* No prior chemotherapy for locally recurrent or metastatic breast cancer.
* At least 12 months since prior adjuvant or neoadjuvant chemotherapy (including prior taxane therapy and prior anti-angiogenic therapy [i.e. bevacizumab or a TKI]).
* No HER-2 -over-expression (3+) breast cancer (unless treated with trastuzumab or lapatinib).
* Subject has measurable disease by RECIST criteria (randomized portion only).
* Eastern Cooperative Oncology Group (ECOG) Performance Score of 0-1.
* Subject must have adequate bone marrow, renal and hepatic function.
* Subject must have PTT < 1.5 x ULN and INR < 1.5.

Exclusion Criteria:

* Subject has received anti-cancer therapy (other than chemotherapy) including investigational agents, or biologic therapy within 21 days or within a period defined by 5 half lives, whichever is shorter, prior to Study Day 1.
* Subject has not recovered to less than or equal to grade 1 clinically significant adverse effects/toxicities of the previous therapy.
* Subject has received radiation therapy within 14 days of Study Day 1.
* Subject has received anti-cancer hormonal therapy within 14 days of Study Day 1.
* Subject has undergone major surgery within 21 days of Study Day 1.
* The subject has untreated brain or meningeal metastases.
* Subject is receiving therapeutic anticoagulation therapy.
* Subject has a history of or currently exhibits clinically significant cancer related events of bleeding (e.g., hemoptysis).
* Subject currently exhibits symptomatic or persistent, uncontrolled hypertension.
* Subject has a history of myocardial infarction, stroke, or transient ischemic attack (TIA) within 6 months of study day 1.
* Subject has a documented left ventricular (LV) ejection fraction < 50%
* Subject has known autoimmune disease with renal involvement.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Radiographic evaluation every 3 months, clincial evaluation monthly

SECONDARY OUTCOMES:
Overall survival | Subject death

CONTACTS AND LOCATIONS:
Overall Officials: Justin L. Ricker, MD, Study Director — AbbVie
Locations (3):
- United States (2):
  - Site Reference ID/Investigator# 8352, San Francisco, California
  - Site Reference ID/Investigator# 6920, Harvey, Illinois
- Site Reference ID/Investigator# 10181, Durango, DGO., Mexico